CLINICAL TRIAL: NCT05512741
Title: Evaluation of the Role of the Intestinal Microbiota in the Mechanism of Postoperative Ileum After Colorectal Surgery : a Preliminary Study
Brief Title: Intestinal Microbiota and Postoperative Ileus After Colorectal Surgery
Acronym: MICRO-IPO
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: MicroIPO2022
Record Dates: First submitted 2022-08-10; First posted 2022-08-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Ileus; Surgery-Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — collection of feces before and after surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group Ileus: Patients that experience POI after colorectal surgery. POI is defined by the presence of 2 of the 5 criteria of Vather from the first postoperative day.
  The first 10 consecutive patients experiencing POI will be included in the study.
  Interventions: Other: Feces collection
- No POI group: Patients that do not experience POI. The 10 patients having the fastest recovery of gastro-intestinal functions after surgery during the period of inclusion will be included in the study
  Interventions: Other: Feces collection

INTERVENTIONS:
Other: Feces collection — Feces will be collected, at home, by the patient., by using a collection kit. The stools are collected in the 2 last days before surgery.
  After surgery, the first stool is collected, during the hospitalization, by using the same kit. Stools are conserved in the same condition, before being frozen in our local biologic ressources center.

SUMMARY:
Postoperative ileus (POI) after colorectal surgery is frequent and is a burden for national health authority because it increases the morbidity and the length of hospital stay.

Some of the stage of the mechanism of POI are known and are now targeted to reduce its occurence but despite these measures, POI still happens in 10-30% of surgeries.

The role of the intestinal microbiota in POI is unknown while it could be a new target to reduce its duration or its occurence.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic colorectal resection with anastomosis and without diverting stoma

Exclusion Criteria:

* risk of modification of the microbiota (terminal enterostomy, chronic inflammatory bowel disease, oesophageal or gastric surgery, vagal nerves lesion, beta lactamin allergy, bowel cleansing)
* postoperative complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with POI and 10 patients without POI selected in the consecutive patients undergoing colorectal surgery during the period of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Composition of the feces microbiota before surgery | within the 2 last days before surgery
  The composition of the microbiota will be assessed by the analysis of the region V3 V4 of the 16S rRNA, amplificateur by high flow sequencing
Composition of the feces microbiota after surgery | up to the first postoperative stools, an average of 3 postoperative days
  The composition of the microbiota will be assessed by the analysis of the region

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, visceral and endocrine surgery department, Angers, France